CLINICAL TRIAL: NCT03298308
Title: Effects of Cranial Electric Stimulation on Brain Wave Activity: A Pilot Study
Brief Title: Brainwave Changes and Cranial Electrotherapy Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 418467-1
Record Dates: First submitted 2017-09-20; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brainwave (Experimental): Brainwave analysis after cranial electric stimulation
  Interventions: Device: Cranial Electric Stimulation

INTERVENTIONS:
Device: Cranial Electric Stimulation — Micro amperage TCDS

SUMMARY:
This pilot study explored relationships between cranial electric stimulation and brainwave changes.

DETAILED DESCRIPTION:
This pilot study will collect data from properly consented and subsequently enrolled subjects in the Psychiatric Continuity Service (PCS). All PCS programs provide both group and individual therapy designed to address various chronic mental health disorders such as major depressive disorder, anxiety, and post-traumatic stress disorder (PTSD). Group therapy and education focus on how chronic mental health disorders develop, the recovery process and psychosocial stressors that may contribute to both improvement in functioning and declines. Every patient is different with regard to how his or her program is tailored, but everyone receives weekly individual counseling from behavioral health providers (psychiatrists, psychologists and clinical social workers). PCS works in tandem with other treatment providers, case managers and chains of command. PCS is also equipped to transfer patients in need to higher levels of care in cases of emergency.

All prospective subjects will be active duty service members who are enrolled in PCS. Subjects will be recruited by the Associate Investigator (AI) or Principal Investigator (PI). The primary outcome measure is the exploration of changes in specific brain wave activity in response to a Cranial Electrotherapy Stimulation (CES) intervention.

Subjects who agree to participate in the study will complete a consent and Health Insurance Portability and Accountability Act (HIPAA) form and baseline questionnaires. In addition, since the fetal effects of the CES device is not known;, female subjects will have to present a negative pregnancy test within one week of the research intervention. Those female subjects to which pregnancy is unlikely (i.e. hysterectomy), will be excluded from a pregnancy test if this information can be verified medically. will self-report regarding as it applies menstrual cycle length and birth control method used within the last two weeks.

The intervention will take place during clinic hours. This will be a one-time intervention that will last approximately 1 to 1 ½ hours. The AI will prepare the CES device, briefly explain the function, and place the CES ear clips on the subject. The CES device will not be turned on at this point. This is similar to clinic practice, however in clinical practice any PCS staff trained in the use of the CES device may prepare and administer the CES device to the patient.

Next the AI will prepare the MindSet EEG device, ensure that it is functioning properly, and obtain signal acquisition. The AI will then explain the brainwave headset (MindSet) to the subject and properly place the headset on their head. Next a series of computer led activities to reduce extraneous artifacts (such as eye blink and muscle movement) will be completed by the subject. Following this, a baseline test measuring brainwave frequencies will be completed by the subject. This will last 30 seconds. Once this is completed, the CES device can be turned on and activated for 20 minutes. The CES micro amperage will be set by the subject based on therapeutic dose and locked in place on the CES device. Immediately following the completion of the 20 minute CES session, an EEG brainwave measure will be completed. Additional brainwave measure will be taken 5 minutes and 10 minutes post the CES session. Each of these brainwave measures will last 30 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria All prospective subjects will be active duty service members who are enrolled in PCS

Exclusion Criteria:

* • Subjects will be excluded who have a seizure disorder, a cardiac pacemaker, or active untreated vertigo.

  * Subjects will be excluded if they have used CES the day of the study. However, they may participate in the study the following day.
  * Female subjects who are or who suspect they may be pregnant.
  * Subjects will also be excluded who are clinically judged by the investigators to be actively suicidal or have another psychiatric condition that would require inpatient hospitalization

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Quantitative EEG Analysis | Quantitative EEG collected at baseline (immediately before stimulation), immediately after 20 minutes of stimulation and then 5 and 10 minutes post stimualtion. Each of these four measures will record 30 seconds of brainwave activity
  The investigators used a commercially available EEG headset (Neurosky MindSet) in combination with EEG software (SmartMind) to obtain and analyze the Quantitative EEG from the subjects. The combination of the EEG headset with the software identified the five brainwave frequencies that are clinically relevant in studying EEG activity: Alpha, Beta, Delta, Gamma, and Theta. The combination of the headset and software reported changes in brainwave amplitude in microvolts for each brainwave frequency. Alpha waves increase with relaxation and drowsiness; and Beta waves, increase with wakefulness and concentration. Delta and Theta waves increase during meditative states and Gamma may suggest brain synchronicity.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lande RG, Gragnani CT. Prospective Study of Brain Wave Changes Associated With Cranial Electrotherapy Stimulation. Prim Care Companion CNS Disord. 2018 Jan 18;20(1):17m02214. doi: 10.4088/PCC.17m02214. PMID 29360291